CLINICAL TRIAL: NCT00453076
Title: Randomized Trial of Conventional Covered Self Expandable Metallic Stent Versus Paclitaxel Eluting Covered Self Expandable Metallic Stent in Unresectable Malignant Bile Duct Obstruction
Brief Title: Paclitaxel Eluting Covered Metallic Stent for Unresectable Malignant Bile Duct Obstruction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Sang Soo Lee, MD, PhD, University of Ulsan College of Medicine, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-11
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2006-11

CONDITIONS: Bile Duct Obstruction
Keywords: Biliary Obstruction
MeSH Terms: conditions — Cholestasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel eluting covered metal stent (Experimental): Paclitaxel eluting covered metal stent group
  Interventions: Device: Paclitaxel eluting covered metal stent and control covered metal stent
- Control covered metal stent (Active Comparator): Control covered metal stent group
  Interventions: Device: Paclitaxel eluting covered metal stent and control covered metal stent

INTERVENTIONS:
Device: Paclitaxel eluting covered metal stent and control covered metal stent — Paclitaxel eluting covered metal stent and control covered metal stent are inserted with standard ERCP technique

SUMMARY:
The primary goal is to determine stent patency and overall survival of the conventional covered self expandable metallic stent versus paclitaxel eluting covered self expandable metallic stent in unresectable malignant bile duct stricture.

The secondary goals are to assess reinterventions, complications, technical difficulties, and physician graded ease of placement and to assess toxicity of paclitaxel eluting covered self expandable metallic stent.

DETAILED DESCRIPTION:
1.1 Self-expandable metallic stent (SEMS) Self-expandable metallic stent (SEMS) placement is a well-established and widely used treatment for patients with unresectable malignant biliary obstruction. This palliative technique prolongs survival, shortens hospital stay, and improves quality of life in patients with unresectable malignant biliary obstruction. Unfortunately, SEMS have the disadvantage of occlusion over time because of tumor ingrowth (tumor invasion through the metal wire mesh of the stent) or overgrowth (tumor growing at the end of the stent), and mucosal hyperplasia as a consequence of chronic irritation. The occlusion rate of SEMS varies from 10% to 50% of cases of malignant biliary obstruction. 6-9 Duration of SEMS patency is important for patients with a short life-expectancy because quality of life and cost-effectiveness are mainly determined by stent occlusion. Previous studies have suggested that covered metallic stents may prevent tumor ingrowth and reduce the occlusion rate, but tumor overgrowth is still problematic. 11 12 13 Therefore, there is a dire need for a metallic stent that prevents both tumor ingrowth and overgrowth.

1.2. Paclitaxel Paclitaxel is a potent antineoplastic drug extracted from the bark of the pacific yew (Taxus brevifolia) and has been utilized for the therapy for ovarian, breast, lung, and other cancers. This potent drug exerts its pharmacological effects through a unique mechanism. Paclitaxel causes formation of numerous decentralized and unorganized microtubules and enhances the assembly of extraordinarily stable and dysfunctional microtubules. In addition, it inhibits activation processes like activation of protein kinases or release of transcription factors. In addition, paclitaxel has several pharmacokinetic characteristics that make it well suited for locoregional cancer therapy. It has rapid cellular uptake and a first pass effect because of its extremely lipophilic character and long lasting action over a broad concentration range. Furthermore, paclitaxel has antiangiogenic and antimetastatic properties. The efficacy in dose dependent inhibition of cell proliferation of human gallbladder epithelial cells, fibroblasts, and pancreatic adenocarcinoma cells makes paclitaxel a very promising substance for local drug delivery to reduce the proliferative and migratory components that are involved in tumor growth. This inhibitory effect of paclitaxel on the cell lines had served as the basis to develop drug-eluting stents for malignant biliary strictures.

1.3. Paclitaxel-eluting covered metallic stent Covering the stent with chemotherapeutic agent, such as paclitaxel, should give protection against tumor ingrowth, overgrowth, or both resulting in increased patency, longer survival rates and increased remaining quality of life. There had been only few studies on the effect of a paclitaxel-eluting covered metallic stent on animal bile duct. In a study on porcine bile duct, the degree of histologic changes, which included inflammatory cell infiltration and fibrous reactions, corresponded to the amount of paclitaxel incorporated within the stent. The degree of inflammatory change was more severe in porcine bile duct in contact with the stent with 20% concentration (% wt/v) of paclitaxel than the stent with 10% concentration. There was no case of transmural necrosis and perforation. The results of this particular study had served as a basis for further research. In our preliminary study, no significant complications such as perforation or stent migration have occurred in either DDS or CS group. Therefore, it can be suggested that this paclitaxel-eluting SEMS is safe in the normal canine bile duct.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable malignancy of the extrahepatic bile duct
* Age >= 18 years and above
* Estimated life expectancy of more than 3 months
* ECOG performance status of 2 or lower
* Adequate bone marrow function
* WBCs > 4,000/µL, absolute neutrophil count [ANC]>1,500/µL
* Hemoglobin >9.0 g/dL
* Platelets > 100,000/µL
* Adequate kidney function (creatinine<1.5 mg/dL)
* No serious medical or psychological condition that would preclude study treatment
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

* Age below 18 years
* Pregnancy
* Active alcohol or drug abuse
* Simultaneously participating in another investigational drug or device study
* Allergy to stainless steel or nitinol
* Allergy to paclitaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-11; Primary Completion 2008-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The primary goal is to determine stent patency and overall survival of the conventional covered self expandable metallic stent versus paclitaxel eluting covered self expandable metallic stent in unresectable malignant bile duct stricture. | Two year

SECONDARY OUTCOMES:
The secondary goals are to assess reinterventions, complications, technical difficulties, and physician graded ease of placement and to assess toxicity of paclitaxel eluting covered self expandable metalic stent. | Two year

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Hwan Kim, MD,PhD, Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea